CLINICAL TRIAL: NCT07047248
Title: Short- and Long-Term Effects of Whole-Body Photobiomodulation in Type II Diabetes Patients: A Protocol for a Controlled Clinical Trial
Acronym: PBM
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Malaga (Other)
Collaborators: clinical professor (Unknown)
Responsible Party: Principal Investigator, Daniel Aguilar Nunez, danunez, University of Malaga
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PBM
Record Dates: First submitted 2025-06-15; First posted 2025-07-02 (Actual); Last update posted 2025-07-02 (Actual); Status verified 2025-06

CONDITIONS: Type II Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: Triple (ParticipantCare ProviderOutcomes Assessor)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention (Experimental): A treatment with whole body red light therapy (NovoTHOR®) will be carried out
  Interventions: Device: PBM
- Placebo (Placebo Comparator): A placebo whole body red light will be carried out
  Interventions: Other: Placebo PBM

INTERVENTIONS:
Device: PBM — A whole body red light therapy (NovoTHOR®) will be carried out during 20 minutes
  Arms: intervention
Other: Placebo PBM — A placebo whole body red light will be carried out during 20 minutes
  Arms: Placebo

SUMMARY:
The development of an integral and global treatment to improve the quality of life in those withType II Diabetes Patients is challenging, thus a whole body Photobiomodulation (PBM) therapy program is proposed as an effective option.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 30 to 70 years.
* Diagnosed with Type 2 Diabetes Mellitus (T2DM) according to the American Diabetes Association (ADA) criteria.
* HbA1c levels between 6.5% and 10% at screening.
* Stable diabetes management regimen (medications and lifestyle) for at least three months prior to enrollment

Exclusion Criteria:

* Presence of severe diabetic complications (e.g., end-stage renal disease, proliferative diabetic retinopathy).
* History of photosensitivity or medical conditions exacerbated by light exposure.
* Use of medications or supplements known to significantly alter glucose metabolism, other than current stable diabetes management.
* Pregnant or lactating women.

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2025-08-30 (Estimated); Primary Completion 2025-09-30 (Estimated); Study Completion 2026-01-30 (Estimated)

PRIMARY OUTCOMES:
Glucose Metabolism: Evaluated through changes in fasting blood glucose levels and HbA1c. | Follow-ups at 3 months and 6 months post-intervention
  • Glucose Metabolism: Evaluated through changes in fasting blood glucose levels and HbA1c.

SECONDARY OUTCOMES:
Sleep Quality: Assessed through the Pittsburgh Sleep Quality Index (PSQI). | Follow-ups at 3 months and 6 months post-intervention
  The Pittsburgh Sleep Quality Index (PSQI) is a widely used self-report questionnaire that assesses sleep quality over a one-month time interval.

CONTACTS AND LOCATIONS:
Locations (1):
- Dr, Granada, Spain